CLINICAL TRIAL: NCT01528891
Title: Dexmedetomidine as a Rapid Bolus for Treatment and Prophylactic Prevention of Emergence Agitation in Anesthetized Children
Brief Title: Dexmedetomidine as a Rapid Bolus in Children for Emergence Agitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peter Davis (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Peter Davis, Anesthesiologist-in-Chief, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO11070498
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Tonsillectomy
Keywords: tonsillectomy; emergence agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- placebo (Placebo Comparator): Normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — 0.5 micrograms/Kilogram one time bolus 5 minutes prior to the end of surgery
  Other Names: Precedex
  Arms: Dexmedetomidine
Other: Placebo
  Arms: placebo

SUMMARY:
To Determine The Efficacy of a Rapid Bolus Injection of Dexmedetomidine on the Incidence of Emergence Agitation in Anesthetized Children and the Cardiovascular Profile of a Rapid Bolus Injection of Dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing tonsillectomy with and without adenoidectomy and myringotomy and tube insertion
* ASA 1,2,3
* females who have started menses but have a negative urine pregnancy test

Exclusion Criteria:

* patients with known dysrhythmias,
* not recovering in the ICU
* developmental delay,
* autism communication disorder
* bleeding disorder
* PI discretion

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 418 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Davis, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 418 patients overall were enrolled in the study. Of these patients, 18 failed screening prior to randomization into either treatment arm.
Groups:
- Dexmedetomidine: Dexmedetomidine
  Dexmedetomidine: 0.5 micrograms/Kilogram one time rapid bolus 5 minutes prior to the end of surgery
- Placebo: Normal saline equivalent volume
  Placebo
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 200 | 200
Completed | 200 | 200
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine: Dexmedetomidine
  Dexmedetomidine: 0.5 micrograms/Kilogram one time rapid bolus 5 minutes prior to the end of surgery
  Of the 200 patients in this treatment arm, 5 were totally excluded from analysis due to administration of medications that were not a part of the anesthetic protocol.
- Placebo: Normal saline equivalent volume
  Placebo
  Of the 200 patients in this treatment arm, 2 were totally excluded from analysis due to administration of medications that were not a part of the anesthetic protocol.
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 195 | 198 | 393
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 195 | 198 | 393
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (1.6) | 5.8 (1.6) | 6.0 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 97 | 193
  Male | 99 | 101 | 200
Region of Enrollment [Number; unit: participants]
  United States | 195 | 198 | 393

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate (HR)
Description: beats per minute (bpm)
Time Frame: Heart rate was measured immediately prior to study drug injection (baseline) and every minute thereafter for 5 minutes. Heart rate was also measured upon the patient's arrival to the Post-Anesthesia Care Unit (PACU).
Population: Heart rate values were compared between groups at each time point and within groups over time.
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Placebo: Normal saline
  Placebo
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 195 | 198
bpm
  Baseline HR | 120 (16) | 121 (16)
  1 min HR | 107 (18) | 121 (16)
  2 min HR | 104 (16) | 120 (15)
  3 min HR | 105 (14) | 119 (15)
  4 min HR | 105 (15) | 118 (15)
  5 min HR | 105 (15) | 117 (15)
  PACU HR | 94 (13) | 108 (16)
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Heart rate values at each time point were compared between groups; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — P<0.01 for the following time points, 1 minute, 2 minutes, 3 minutes, 4 minutes, 5 minutes, and PACU. P-values are adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Dexmedetomidine; Heart rate values were compared over time against the baseline value; Test type: Superiority or Other; p < 0.01, ANOVA — P<0.01 for the following time points, as compared to the baseline value: 1 minute, 2 minutes, 3 minutes, 4 minutes, 5 minutes, and PACU. P-values are adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Placebo; Heart rate values were compared over time against the baseline value; Test type: Superiority or Other; p < 0.01, ANOVA — P<0.01 for the following time points, as compared to the baseline value: 4 minutes, 5 minutes, and PACU. P-values are adjusted for multiple comparisons

2. Secondary Outcome: Incidence of Emergence Agitation (EA)
Description: Using a Pediatric Anesthesia Emergence Delirium (PAED) score, emergence agitation scores will be recorded. The PAED score consists of 5 different criteria which are assessed from 0 to 4 once the patient has woken up. These criteria are then totaled; the total may range from 0 to 20, where 0 represents no emergence agitation and 20 represents maximal agitation. For this study, patients with a maximum PAED score of >10 and >12 were considered to be agitated.
Time Frame: The highest PAED score for each patient within the first 30 minutes after waking up was recorded.
Population: There were 2 patients in the Dexmedetomidine group and 9 patients in the placebo group who were excluded from analysis of emergence agitation. These patients were excluded because they received medications that were not a part of the anesthetic protocol and could affect their PAED score.
Measure: Number; unit: percentage of patients with EA
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 193 | 189
percentage of patients with EA
  EA using PAED >10 threshold | 36 | 66
  EA using PAED >12 threshold | 30 | 61
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; The incidence of agitated patients in each group was compared; Test type: Superiority or Other; p < 0.0001, Fisher Exact — P<0.0001 was calculated for both groups

3. Primary Outcome: Systolic Blood Pressure (SBP)
Description: mmHg
  Two subjects with missing data points for SBP were necessarily eliminated from repeated measures analysis.
Time Frame: Systolic blood pressure (SBP) was measured immediately prior to study drug injection (baseline) and every minute thereafter for 5 minutes. SBP was also measured upon the patient's arrival to the Post-Anesthesia Care Unit (PACU).
Population: Systolic blood pressure values were compared between groups at each time point and within groups over time.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 194 | 197
mmHg
  Baseline SBP | 99 (16) | 99 (16)
  1 min SBP | 104 (16) | 100 (15)
  2 min SBP | 99 (14) | 99 (14)
  3 min SBP | 95 (13) | 98 (14)
  4 min SBP | 93 (13) | 97 (15)
  5 min SBP | 92 (13) | 96 (15)
  PACU SBP | 97 (12) | 105 (17)
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Systolic blood pressure values were compared between groups at each time point; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — P<0.01 for the following time points: 1 minute, 4 minutes, 5 minutes, and PACU. P-values are adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Dexmedetomidine; SBP values were compared against the baseline value within each group over time; Test type: Superiority or Other; p < 0.01, ANOVA — P<0.01 for the following time points, as compared to the baseline value: 1 minute, 3 minutes, 4 minutes, and 5 minutes. P-values are adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Placebo; SBP values were compared against the baseline within each group over time; Test type: Superiority or Other; p < 0.01, ANOVA — P<0.01 for the following time points, as compared to the baseline value: 5 minutes and PACU. P-values were adjusted for multiple comparisons

4. Primary Outcome: Diastolic Blood Pressure (DBP)
Description: mmHg
  Three subjects with missing data points for DBP were necessarily eliminated from repeated measures analysis.
Time Frame: Diastolic blood pressure (DBP) was measured immediately prior to study drug injection (baseline) and every minute thereafter for 5 minutes. DBP was also measured upon the patient's arrival to the Post-Anesthesia Care Unit (PACU).
Population: Diastolic blood pressure values were compared between groups at each time point and within groups over time.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 194 | 196
mmHg
  Baseline DBP | 47 (9) | 47 (9)
  1 min DBP | 52 (10) | 47 (9)
  2 min DBP | 48 (9) | 47 (8)
  3 min DBP | 45 (8) | 46 (8)
  4 min DBP | 44 (8) | 45 (9)
  5 min DBP | 43 (8) | 45 (8)
  PACU DBP | 50 (7) | 55 (11)
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; DBP values were compared between groups at each time point; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — P<0.01 for the following time points: 1 minute and PACU. P-values were adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Dexmedetomidine; DBP values were compared within each group against the baseline value; Test type: Superiority or Other; p < 0.01, ANOVA — P<0.01 for the following time points, as compared to baseline: 1 minute, 3 minutes, 4 minutes, 5 minutes, PACU. P-values were adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Placebo; DBP values were compared against the baseline value within each group over time; Test type: Superiority or Other; p < 0.01, ANOVA — P<0.01 for the following time points, as compared to baseline: 4 minutes, 5 minutes, PACU. P-values were adjusted for multiple comparisons

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/200 | 0/200
Other Adverse Events (participants affected / at risk) | 18/200 | 34/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=200) | Placebo (N=200)
Desaturation with Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — The serious adverse event (SAE) was associated with a prolonged hospital stay. The investigators felt the SAE was unrelated to the study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=200) | Placebo (N=200)
Dizziness (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2)
Congestion (General disorders) | 3 (3) | 0 (0)
Bronchospasm (General disorders) | 0 (0) | 1 (1)
Laryngospasm (General disorders) | 0 (0) | 7 (7)
Tachypnea (General disorders) | 1 (1) | 0 (0)
Stridor (General disorders) | 1 (1) | 3 (3)
Hypercapnia (General disorders) | 0 (0) | 1 (1)
Apnea (General disorders) | 1 (1) | 0 (0)
Emesis (General disorders) | 3 (3) | 2 (2)
Croupy Cough (General disorders) | 1 (1) | 3 (3)
Desaturation (General disorders) | 1 (1) | 5 (5)
Enuresis (General disorders) | 2 (2) | 1 (1)
Bigeminal Premature Atrial Contractions (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 3 (3)
Rigor (General disorders) | 0 (0) | 1 (1)
Wheezing (General disorders) | 0 (0) | 1 (1)
Pruritus (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Excess Secretions (General disorders) | 0 (0) | 1 (1)
Intravenous Infiltration (General disorders) | 0 (0) | 1 (1)
Bleeding (General disorders) | 4 (4) | 9 (9)
Kinked intravenous catheter (General disorders) | 1 (1) | 0 (0)
Poor oral intake (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No